CLINICAL TRIAL: NCT03924128
Title: Study of the Effects of Photobiomodulation in Patients With Osteoarthritis
Status: No longer available | Type: Expanded Access
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, marucia chacur, PhD, University of Sao Paulo
Other Study IDs: 93744418.5.0000.0068
Record Dates: First submitted 2019-04-17; First posted 2019-04-23 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-10

CONDITIONS: Osteo Arthritis Knee; Pain, Chronic; Inflammation
MeSH Terms: conditions — Chronic Pain; Inflammation | interventions — Low-Level Light Therapy

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Device: Photobiomodulation — The Photobiomodulation device should cover the entire knee junction, with time of application from 6 to 8 minutes and device turned on.

SUMMARY:
PhotoBioModulation (PBM) is a mature science with therapeutic efficacy in humans and animals, and with excellent results in different medical specialties without side effects. However there are gaps that prevent adoption on a large scale. Recent research developed by our group and partners allowed us to understand the mechanisms of action of PBM, from Molecular Physics through Biochemistry and with consequent clinical validation, with precise, replicable and personalized therapeutic results. These findings have led to treatments for many kinds of pains with industrial predictability and accuracy, phenotypic adequacy technologies that are encapsulated, prescribed, and applied. Photobiomodulation applications cover treatments for pain, inflammation, tissue regeneration, healing, immune system activation, all of which are essential characteristics for osteoarthritis therapy. Our idea is to formulate great challenges of Photobiomodulation as a solution to osteoarthritis as follows: 1) Make PBM-based therapies as predictable as drug-based therapies; this is possible with precise dose calculation performed by our team; 2) Map the biochemical and molecular effects of PBM, including those related to gene expression; 3) Unify PBM theory by synthesizing and giving meaning to the millions of PBM data associated with osteoarthritis and correlating with clinical study to be performed under this thematic project. Overcoming these challenges, PBM will become a complementary (or supplementary) alternative to medications, physiotherapy and surgical procedures for the treatment of osteoarthritis.

DETAILED DESCRIPTION:
Treatment Procedure Treatment was administered twice a week on the same days over a period of 5 weeks with the system Light-Aid (Bright Photomedicine, SP, Brazil), operated at continuous wave, with 100 LED of 850 nm wavelength) or with a placebo probe of same appearance and display. The irradiation parameters were customized based on the disease, pain intensity, skin phototype and BMI. The probes were numbered A (active) and B (placebo). Treatment was administered in contact to the skin over the patient's knee. Both knees were treated but statistical analysis was done only for the worst one.

Knee Pain scores Visual analogue scale (VAS) was used to evaluate pain. Patients were instructed to number their level of pain from 0 (absence of pain) to 10 (worst possible pain). The VAS was applied after each PBMT session, and weekly for sixteen weeks after treatment Quality of life Two Quality of Life (QOL) questionnaires were used: Knee injury and Osteoarthritis Outcome Score (KOOS) and World Health Organization Quality of Life-bref (WHOQOL-abbreviated). Both evaluations were recorded and compared before and after the last session of treatment.

The KOOS evaluate both short-term and long-term consequences of knee injury and OA. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related QOL. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.

The WHOQOL assesses the individual's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns. The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment.

Physical Function For functional assessments, the timed up and go test (TUG) and the sit-to-stand test (STS) were used. TUG determines fall risk and measures the progress of balance, sit to stand and walking. STS test is a method for lower extremity strength assessment. Both evaluations were recorded and compared before and after the last treatment session and the details of it can be found in supplementary material.

For the TUG and STS, patients were instructed to initiate the test at a sitting position, with the trunk in an erect posture, arms crossed over the chest, and feet on the floor. TUG is a mobility test that evaluates the time that the patient takes to get up from a chair, walk a distance of 3 m at a normal speed until he/she reaches a mark on the ground, then turn around, walk back and sit on the chair without the support of the arms. Patients were instructed to perform the sit-to-stand movements as fast as possible in 30 seconds. The number of completed sit-to-stands in 30 seconds was recorded.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age ≥ 20 years old
* Diagnosed with Osteoarthritis stages III and IV according to the American College of Rheumatology
* Pain
* Functional impairment for more than 3 months, able to wander with or without canes.

Exclusion Criteria:

* History of cancer
* Unstable cardiovascular disease
* uncontrolled hypertension
* morbid obesity, that is, BMI ≥ 40
* terminal illness
* cerebrovascular disease
* dementia
* heart pacemaker
* superior or inferior limb fractures.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Nathalia Lopes Ferreira, graduate, Principal Investigator — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil